CLINICAL TRIAL: NCT05919082
Title: A Phase 3, Randomised, Investigator-blind, Active-controlled, Parallel Group, Multicentre Trial Comparing the Efficacy and Safety of 4-weeks Treatment With LEO 90100 and Daivobet® Ointment in Adult Chinese Subjects With Stable Plaque Psoriasis
Brief Title: A Study to Investigate Efficacy and Safety With LEO 90100 Compared With Daivobet® Ointment in Adult Chinese Subjects With Stable Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LP0053-2277; U1111-1285-7764 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Stable Plaque Psoriasis
Keywords: Stable plaque psoriasis; Vitamin D analogue; Native Chinese subjects

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LEO 90100 (Experimental): The subjects will receive LEO 90100 foam once daily for 4 weeks.
  Interventions: Drug: LEO 90100
- Daivobet® ointment (Active Comparator): The subjects will receive Daivobet® ointment once daily for 4 weeks.
  Interventions: Drug: Daivobet® ointment

INTERVENTIONS:
Drug: LEO 90100 — Subjects will apply LEO 90100 topically; up to 15 g per day (or 105 g per week).
  Arms: LEO 90100
Drug: Daivobet® ointment — Subjects will apply Daivobet® ointment topically; up to 15 g per day (or 105 g per week).
  Arms: Daivobet® ointment

SUMMARY:
This study is conducted to assess the efficacy and safety of LEO 90100 when used on the body for the treatment of stable plaque psoriasis in native adult Chinese subjects, compared to Daivobet® ointment.

DETAILED DESCRIPTION:
This study is phase 3, randomised, prospective, investigator-blinded, active-controlled, parallel group, multicentre trial to evaluate the efficacy and safety of 4 weeks treatment with LEO 90100 compared with Daivobet® ointment. Eligible participants will be randomised in a 1:1 ratio to either LEO 90100 or Daivobet® ointment treatment.

The trial will last for 6 weeks to 10 weeks for each participant, which includes wash out period and treatment period of up to 4 weeks and a safety follow up period of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chinese native
* Aged 18 or over
* A clinical diagnosis of stable plaque psoriasis for at least 6 months
* Stable plaque psoriasis on the trunk and/or limbs (excluding psoriasis on the face, scalp, genitals, and skin folds) involving 2-30% of the body surface at Day 1 (Visit 2) of the trial.
* Having a Physician Global Assessment of at least 'mild' at Day 1 (Visit 2)
* An mPASI score of at least 2 on the trunk and/or limbs at Day 1 (Visit 2)
* Women of childbearing potential must use an adequate form of birth control throughout the trial and for at least 8 weeks after last administration of IMP
* Male subjects with a female partner of childbearing potential must use adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice)
* Having a signed and dated informed consent.

Exclusion Criteria:

* Systemic use of biological treatments with a potential effect on psoriasis vulgaris within the specified time periods prior to treatment assignment (depending on treatment)
* Systemic treatments with all therapies other than biological treatments with a potential effect on psoriasis vulgaris within 4 weeks prior to treatment assignment
* Psoralen combined with ultraviolet A therapy (PUVA) within 4 weeks prior to treatment assignment
* Systemic treatment with Apremilast within 4 weeks prior to treatment assignment
* Ultraviolet B (UVB) therapy within 2 weeks prior to treatment assignment
* Topical treatment of psoriasis with strong corticosteroids within 2 weeks prior to treatment assignment
* Topical treatment of psoriasis with traditional Chinese medicine within 2 weeks prior to treatment assignment
* Treatment with any non-marketed drug substance (any agent which has not yet been made available for clinical use) within 4 weeks/5 half-lives prior to treatment assignment
* Any other topical treatment that could affect plaque psoriasis within 2 weeks prior to treatment assignment
* Current diagnosis of guttate, erythrodermic, exfoliative, pustular or unstable psoriasis
* Patients with any of the following conditions present on any skin area: viral lesions, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, acne vulgaris, acne rosacea, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, ulcers and wounds
* Disorders of calcium metabolism
* Renal insufficiency, hepatic disorders or severe heart disease
* Cushing's disease or Addison's disease
* Known or suspected hypersensitivity to any component(s) of the investigational medicinal product (IMP)
* Current participation in any other interventional clinical trial
* Previously screened in this trial
* Participation in another clinical trial within 4 weeks prior to treatment assignment
* Women who are pregnant, wishing to become pregnant or are breast-feeding
* Chronic alcohol or drug abuse within 12 months prior to screening, or any condition associated with poor compliance
* Employees of the trial site or any other individuals directly involved with the planning or conduct of the trial, or immediate family members of such individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (29):
- China (29):
  - LEO Pharma Investigational Site, Bengbu, Anhui
  - LEO Pharma Investigational Site, Hefei, Anhui
  - LEO Pharma Investigational Site, Beijing, Beijing Municipality
  - LEO Pharma Investigational Site, Chongqing, Chongqing Municipality
  - LEO Pharma Investigational Site, Guangzhou, Guangdong
  - LEO Pharma Investigational Site, Shenzhen, Guangdong
  - LEO Pharma Investigational Site, Cangzhou, Hebei
  - LEO Pharma Investigational Site, Chengde, Hebei
  - LEO Pharma Investigational Site, Shijiangzhuang, Hebei
  - LEO Pharma Investigational Site, Nanyang, Henan
  - LEO Pharma Investigational Site, Shiyan, Hubei
  - LEO Pharma Investigational Site, Wuhan, Hubei
  - LEO Pharma Investigational Site, Changsha, Hunan
  - LEO Pharma Investigational Site, Baotou, Inner Mongolia
  - LEO Pharma Investigational Site, Hohhot, Inner Mongolia
  - LEO Pharma Investigational Site, Wuxi, Jiangsu
  - LEO Pharma Investigational Site, Yangzhou, Jiangsu
  - LEO Pharma Investigational Site, Zhenjiang, Jiangsu
  - LEO Pharma Investigational Site, Changchun, Jilin
  - LEO Pharma Investigational Site, Xi'an, Shaanxi
  - LEO Pharma Investigational Site, Dongying, Shandong
  - LEO Pharma Investigational Site, Jinan, Shandong
  - LEO Pharma Investigational Site, Shanghai, Shanghai Municipality
  - LEO Pharma Investigational Site, Chengdu, Sichuan
  - LEO Pharma Investigational Site, Suining, Sichuan
  - LEO Pharma Investigational Site, Hangzhou, Zhejiang
  - LEO Pharma Investigational Site, Jiaxing, Zhejiang
  - LEO Pharma Investigational Site, Ningbo, Zhejiang
  - LEO Pharma Investigational Site, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 39 sites that enrolled participants in China from 21 June 2023 to 05 March 2024.
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- LEO 90100: The participants received up to 15 g LEO 90100 foam once daily for 4 weeks.
- Daivobet Ointment: The participants received up to 15 g Daivobet® ointment once daily for 4 weeks.
Period: Overall Study
Arm/Group | LEO 90100 | Daivobet Ointment
Started | 302 | 302
Completed | 290 | 291
Not Completed | 12 | 11
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Lack of Efficacy | 0 | 1
Not completed — Investigator Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 90100 | Daivobet Ointment | Total
Number analyzed (Participants) | 302 | 302 | 604
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (13.45) | 45.7 (13.07) | 45.8 (13.25)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 3 | 3
  Between 18 and 65 years | 273 | 276 | 549
  >=65 years | 29 | 23 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 88 | 166
  Male | 224 | 214 | 438
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 302 | 302 | 604

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Physician's Global Assessment of Disease Severity (PGA) Score of 0 (Clear) or 1 (Almost Clear) at Day 29, With at Least a 2-point Reduction From Baseline
Description: The efficacy of LEO 90100 compared with Daivobet® ointment on severity and extent of stable plaque psoriasis was evaluated.
  The PGA is an instrument used in clinical trials to rate the severity of psoriasis. It is a 5-point scale measurement ranging from 0 to 4, where 0- clear, 1- almost clear, 2- mild, 3- moderate and 4- severe; based on degree of plaque thickening, scaling and erythema. Higher score showed worse outcome.
Time Frame: On Day 29
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Daivobet® Ointment: The participants received up to 15 g Daivobet® ointment once daily for 4 weeks.
Arm/Group | LEO 90100 | Daivobet® Ointment
Number analyzed (Participants) | 302 | 302
Percentage of Participants | 50.0 [44.36 to 55.64] | 42.4 [36.81 to 47.96]
Statistical Analysis 1: Comparison: LEO 90100 vs Daivobet® Ointment; Test type: Other; p = 0.0438, Regression, Logistic; Odds Ratio (OR) = 1.4, 95% CI 2-sided [1.01 to 1.99] — The odds ratio and p-value are obtained by logistic regression model, adjusted for baseline PGA. Wald CI was presented

2. Secondary Outcome: Percentage of Participants With Decrease in Modified Psoriasis Area and Severity Index of at Least 75% (mPASI-75) From Baseline to Day 29
Description: The efficacy of LEO 90100 compared with Daivobet® ointment on severity and extent of stable plaque psoriasis was evaluated.
  The extent of psoriatic involvement will be recorded for each of the areas (trunk [including the neck] and the limbs [such as arms and legs]; excluding any involvement on face, scalp, genitals and skin folds) using the following scale: 0=no involvement, 1=< 10%, 2=10%-29%, 3=30%-49%, 4=50%-69%, 5=70%-89%, 6=90%-100%. The severity of the psoriatic lesions in each of the areas will be recorded for each of the clinical signs of redness, thickness and scaliness. Each clinical sign is scored on a scale of 0-4, reflecting the average severity of all psoriatic lesions on the given body region. Higher score indicates more severity. The overall mPASI can range from 0 to 64.8.
Time Frame: From Baseline to Day 29
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LEO 90100 | Daivobet® Ointment
Number analyzed (Participants) | 302 | 302
Percentage of Participants | 63.6 [58.15 to 69.00] | 53.6 [48.02 to 59.27]
Statistical Analysis 1: Comparison: LEO 90100 vs Daivobet® Ointment; Test type: Other; p = 0.0108, Regression, Logistic; Odds Ratio (OR) = 1.5, 95% CI 2-sided [1.10 to 2.12] — The odds ratio and p-value were obtained by logistic regression model, adjusted for baseline PGA and baseline mPASI score. Wald CI was presented

3. Secondary Outcome: Percentage of Participants With Decrease in mPASI of at Least 90% (mPASI-90) From Baseline to Day 29
Description: as for outcome 2
Time Frame: From Baseline to Day 29
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LEO 90100 | Daivobet® Ointment
Number analyzed (Participants) | 302 | 302
Percentage of Participants | 33.1 [27.80 to 38.42] | 24.5 [19.65 to 29.35]
Statistical Analysis 1: Comparison: LEO 90100 vs Daivobet® Ointment; Test type: Other; p = 0.0199, Regression, Logistic; Odds Ratio (OR) = 1.5, 95% CI 2-sided [1.07 to 2.19] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: The safety of LEO 90100 compared with Daivobet® ointment treating stable plaque psoriasis was evaluated.
  Only treatment emergent adverse events (TEAEs) have been reported for this outcome measure.
  An event was considered treatment-emergent if it started after the first investigational medicinal product (IMP) administration or if it started before the first IMP administration and worsened in severity after the first IMP administration.
Time Frame: From Baseline to Day 43
Population: All participants who are exposed to the IMP. Participants were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100 | Daivobet Ointment
Number analyzed (Participants) | 300 | 301
Participants
  Any TEAE | 77 | 68
  Leading to Deaths | 0 | 0
  Serious | 4 | 0
  Non-Serious | 75 | 68
  Leading to Permanent Discontinuation from investigational medicinal product (IMP) | 3 | 0
  Leading to Withdrawals from the Trial | 3 | 0

ADVERSE EVENTS:
Time Frame: Up to 10 weeks in total
Description: All participants who were exposed to the IMP. Participants were analyzed according to the treatment they actually received.
  All the TEAEs that were accounted throughout the study have been included in this section.
Arm/Group | LEO 90100 | Daivobet Ointment
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/301
Serious Adverse Events (participants affected / at risk) | 4/300 | 0/301
Other Adverse Events (participants affected / at risk) | 53/300 | 39/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 (N=300) | Daivobet Ointment (N=301)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 (N=300) | Daivobet Ointment (N=301)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 18 (18)
Folliculitis (Infections and infestations) | 7 (7) | 4 (4)
Tinea versicolour (Infections and infestations) | 4 (4) | 3 (3)
Fungal infection (Infections and infestations) | 3 (3) | 0 (0)
Cortisol decreased (Investigations) | 7 (7) | 6 (6)
Urine calcium/creatinine ratio increased (Investigations) | 6 (6) | 5 (5)
Application site pain (General disorders) | 3 (3) | 1 (1)
Application site pruritus (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Application site paraesthesia (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 12 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 12 months, the investigator has the right to publish the results from clinical trial generated by him/herself.

DOCUMENTS (2):
  • Study Protocol (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT05919082/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT05919082/SAP_001.pdf